CLINICAL TRIAL: NCT00659724
Title: The Gambro Polyflux HD-C4 Big Ease Of Use And Thrombogenicity Study
Brief Title: Ease of Use and Blood Clotting for the Gambro Polyflux HD-C4 Big Dialyzer
Status: Completed | Type: Observational
Sponsor: Vantive Health LLC (Industry)
Collaborators: Advanced Dialysis Center of Potomac (Industry); Advanced Dialysis Center of Easton (Industry); Gambro Renal Products, Inc. (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Gambro 1462
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Failure
Keywords: Dialyzer
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect information on the ease of use and thrombogenicity of the Polyflux HD-C4 Big and Fresenius Optiflux 180NR or 200NR dialyzers under conditions of routine clinical use for hemodialysis.

DETAILED DESCRIPTION:
This ease of use study involves the use of FDA 510(k) cleared hemodialyzers and will have no impact on the patient's routine dialysis therapy. This study is aimed at obtaining feedback from the nursing and technical staff regarding the use and thrombogenicity of the Polyflux HD-C4 Big, and Fresenius Optiflux 180NR or 200NR dialyzers. The dialysis nursing staff will complete ease of use and thrombogenicity assessments following routine dialysis therapy. Any adverse events will be tracked for the study patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients 18 years of age or older

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Assessment of dialyzer ease of use and thrombogenicity assessments following routine dialysis therapy of 33 adult patients (18 years of age or older)
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Advanced Dialysis Center of Easton, Easton, Maryland
  - Advanced Dialysis Center of Potomac, Arlington, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Hemodialysis Patients: Hemodialysis patients 18 years of age or older receiving routine dialysis treatment for chronic renal failure.
Period: Weeks 1-2: Assessment of 180NR or 200NR
Arm/Group | Hemodialysis Patients
Started | 33
Completed | 33
Not Completed | 0
Period: Weeks 3-4: Assessment of HD-C4 Big
Arm/Group | Hemodialysis Patients
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hemodialysis Patients
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 15
Height [Mean (Standard Deviation); unit: inches] | 65.6 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Ease of Use: Priming Blood Side
Description: For every study treatment/dialyzer, the nursing staff rated the ease of priming blood side as follows:
  Very Easy:Air is easily removed without knocking or clamping procedures. Acceptable:Knocking and/or clamping required for efficient air removal. Difficult:Knocking and/or clamping and additional volume of saline or extended recirculation needed to remove air.
  Very Difficult:Air could not be removed.
Time Frame: Priming at each treatment
Measure: Number; unit: Number of Dialyzers
Units Other Than Participants: Dialyzers
Arm/Group | Revaclear MAX | Optiflux F180NR | Optiflux F200NR
Number analyzed (Participants) | 33 | 33 | 33
Number analyzed (Dialyzers) | 219 | 95 | 97
Number of Dialyzers
  Very Easy | 139 | 13 | 13
  Acceptable | 80 | 82 | 84

2. Primary Outcome: Ease of Use: Priming Dialysate Side
Description: For every study treatment/dialyzer, the nursing staff rated the ease of priming dialysate side as follows:
  Dialysate Side at 500 ml Priming Volume (check one):
  Perfect: No air visible. Acceptable: Some air visible, but considered insignificant. Not Acceptable: Additional actions needed to sufficiently remove air.
Time Frame: Priming at each treatment
Measure: Number; unit: Number of Dialyzers
Units Other Than Participants: Dialyzers
Arm/Group | Revaclear MAX | Optiflux F180NR | Optiflux F200NR
Number analyzed (Participants) | 33 | 33 | 33
Number analyzed (Dialyzers) | 220 | 95 | 97
Number of Dialyzers
  Perfect | 131 | 4 | 2
  Acceptable | 89 | 91 | 95

3. Primary Outcome: Dialyzer Assessment: Fiber Condition
Description: For every study treatment/dialyzer, the nursing staff rated the condition of the dialyzer fibers after rinse-back as follows:
  Very Good:All fibers appear white. Good:Few fibers (less than 10) appear PINK / RED. (check one) Poor:Several fibers (more than 10) appear PINK / RED. (check one) Very Poor:Most fibers (more than 75%) appear PINK / RED. (check one)
Time Frame: Each treatment: assessment of the condition of the dialyzer fibers after rinse-back
Measure: Number; unit: Number of Dialyzers
Units Other Than Participants: Dialyzers
Arm/Group | Revaclear MAX | Optiflux F180NR | Optiflux F200NR
Number analyzed (Participants) | 33 | 33 | 33
Number analyzed (Dialyzers) | 218 | 95 | 97
Number of Dialyzers
  Very Good | 126 | 23 | 15
  Good | 75 | 44 | 45
  Poor | 12 | 17 | 30
  Very Poor | 5 | 11 | 7

4. Primary Outcome: Dialyzer Assessment: Arterial Header Condition
Description: For every study treatment/dialyzer, the nursing staff rated the condition of the arterial header after rinse-back as follows:
  Very Good:Surface as clean as expected. Good:Distinct red ring appears at the dialyzer wall. Poor:Significant appearance of clots, randomly distributed on the surface. Very Poor:Completely red and/or covered with clots.
Time Frame: Each treatment: assessment of the condition of the arterial header after rinse-back
Measure: Number; unit: Number of Dialyzers
Units Other Than Participants: Dialyzers
Arm/Group | Revaclear MAX | Optiflux F180NR | Optiflux F200NR
Number analyzed (Participants) | 33 | 33 | 33
Number analyzed (Dialyzers) | 218 | 95 | 96
Number of Dialyzers
  Very Good | 155 | 0 | 0
  Good | 49 | 66 | 64
  Poor | 13 | 26 | 30
  Very Poor | 1 | 3 | 2

5. Primary Outcome: Dialyzer Assessment: Venous Header Condition
Description: For every study treatment/dialyzer, the nursing staff rated the condition of the venous header after rinse-back as follows:
  Very Good:Surface as clean as expected. Good:Distinct red ring appears at the dialyzer wall. Poor:Significant appearance of clots, randomly distributed on the surface. Very Poor:Completely red and/or covered with clots.
Time Frame: Each treatment: the assessment of the condition of the venous header after rinse-back
Measure: Number; unit: Number of Dialyzers
Units Other Than Participants: Dialyzers
Arm/Group | Revaclear MAX | Optiflux F180NR | Optiflux F200NR
Number analyzed (Participants) | 33 | 33 | 33
Number analyzed (Dialyzers) | 217 | 94 | 97
Number of Dialyzers
  Very Good | 65 | 0 | 0
  Good | 140 | 31 | 35
  Poor | 7 | 52 | 57
  Very Poor | 5 | 11 | 5

ADVERSE EVENTS:
Arm/Group | Hemodialysis Patients
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No